CLINICAL TRIAL: NCT02160990
Title: Effect of Exenatide in Obese Patients With Accelerated Gastric Emptying
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Michael Camilleri, Primary Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-002683 Exenatide; R01DK067071 (NIH); UL1TR000135 (NIH)
Record Dates: First submitted 2014-06-04; First posted 2014-06-11 (Estimated); Results first posted 2016-08-09 (Estimated); Last update posted 2016-08-09 (Estimated); Status verified 2016-06

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity | interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exenatide (Experimental): Participants randomized to this arm received 5 mcg exenatide subcutaneously twice daily for 30 days.
  Interventions: Drug: Exenatide
- Placebo (Placebo Comparator): Participants randomized to this arm received placebo subcutaneously twice daily for 30 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Exenatide — 5 mcg exenatide subcutaneously twice daily for 30 days
  Other Names: Byetta
  Arms: Exenatide
Drug: Placebo — placebo subcutaneously twice daily for 30 days
  Arms: Placebo

SUMMARY:
The overall goal of this study was to determine the effect of exenatide on gastric emptying, satiety and satiation in obese participants. The hypothesis in this study was that exenatide retards gastric emptying in obese patients with baseline accelerated gastric emptying.

DETAILED DESCRIPTION:
This study evaluated the effect of exenatide 5mcg subcutaneous (SQ) twice daily for 30-days versus placebo on gastric emptying, satiety, satiation and weight loss in obese participants with documented accelerated gastric emptying of solids.

Visit 1: Screening - physical exam, questionnaires, pregnancy test. Participants were instructed to continue on the same diet and exercise routine during the entire study.

Visit 2: Satiation Study Day - Subjects returned to the clinic after after fasting for at least 8 hours. A baseline satiation/nutrient drink test was performed on Day 0 prior to initiation of exenatide or placebo. The satiation/nutrient drink test involved drinking a liquid meal (Ensure) at a rate of one ounce per minute until no more could be ingested. At the same time, subject's symptoms were recorded while they drank the liquid meal and for 30 minutes after they reached the maximum volume tolerated. Subjects were randomized to exenatide or placebo, then received 30 days' supply of blinded study medication.

Visit 3: Satiation Study Day - (This test was performed in the last 5 days of the 30 days of medication administration.) Subjects returned to the clinic after after fasting for at least 8 hours. Subjects were instructed to inject exenatide or placebo 30 minutes before the start of the satiation/nutrient drink test. The satiation/nutrient drink test was repeated.

Visit 4: Gastric Emptying by Scintigraphy Day - (This test was performed in the last 5 days of the 30 days of medication administration.) Subjects returned to the clinic after after fasting for at least 8 hours. Subjects were instructed to inject exenatide or placebo 30 minutes before the start of the gastric emptying test. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs contain a small amount of radioactive substance. At the completion of the breakfast test meal, subjects were instructed to stand in front of a special camera and pictures were taken at specific intervals. On the same day, subjects participated in an all you can eat meal. This meal consists of lasagna, pudding, and skim milk. Food containers were weighed after the meal and calories consumed were estimated using validated dietary software.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects with BMI> 30 Kg/m^2: Otherwise healthy individuals who are not currently on treatment for cardiac, pulmonary, gastrointestinal, hepatic, renal, hematological, neurological, endocrine (other than hyperglycemia not requiring medical therapy) and unstable psychiatric disease.
* Women of childbearing potential will have negative pregnancy test before initiation of medication.
* Gastric emptying (GE): Accelerated GE T1/2 < 79 minutes or GE 1h>35 %

Exclusion Criteria:

* Type 1 or type 2 diabetes mellitus diagnosed according to American Diabetes Association criteria
* Unstable heart disease as evidenced by ongoing angina
* Congestive heart failure
* Concomitant use of appetite suppressants (i.e., caffeine based or diethylpropion) or orlistat (Xenical®)
* Uncontrolled hypertension (Blood pressure greater than 160/90 mmHg)
* Use of anti-diabetic drugs including metformin,
* History of nephrolithiasis,
* Recurrent major depression, presence or history of suicidal behavior or ideation with intent to act, and current substantial depressive symptoms (Patient Health Questionnaire (PHQ-9) total score ≥10).
* Gastroparesis
* Inflammatory bowel disease or irritable bowel syndrome
* Malignancy treated with chemotherapy within the past 3 years
* History of pancreatitis
* Renal insufficiency (eGFR less than 50 ml/min)
* Concomitant use of monoamine oxidase inhibitors (i.e., phenelzine, selegiline), serotonergic agents, and other centrally acting appetite suppressants
* Significant psychiatric dysfunction based upon screening with the Hospital Anxiety and Depression Scale (HADS) self-administered alcoholism screening test (SAAST, substance abuse) and the questionnaire on eating and weight patterns (binge eating disorders and bulimia). If such a dysfunction is identified by a HADS score ≥11 in any of the subscales or difficulties with substance or eating disorders, the participant will be excluded and given a referral letter to his/her primary care doctor for further appraisal and follow-up.
* Intake of medication that could interfere with the interpretation of the study or cause drug interaction (i.e., ketoconazole, erythromycin). Specifically, birth control pill, estrogen replacement therapy, and thyroxine replacement are permissible.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Acosta A, Camilleri M, Burton D, O'Neill J, Eckert D, Carlson P, Zinsmeister AR. Exenatide in obesity with accelerated gastric emptying: a randomized, pharmacodynamics study. Physiol Rep. 2015 Nov;3(11):e12610. doi: 10.14814/phy2.12610. PMID 26542264

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Exenatide | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [33 to 46.8] | 42.5 [25.3 to 49.5] | 39.3 [25.3 to 49.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Gastric Emptying Half-time (T 1/2) of Solids
Description: Gastric emptying of solids half-time is defined as the time for half of the ingested solids to leave the stomach. Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs contained a small amount of a radioactive substance. Anterior and posterior gamma camera images were obtain immediately after radiolabeled meal ingestion, every 15 minutes for the first 2 hours, then 30 minutes for the next 2 hours (total 4 hours after the radiolabeled meal).
Time Frame: time frame is 30 days after the initiation of dose.
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
minutes | 187 [141 to 240] | 86 [73 to 125]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA

2. Secondary Outcome: Percentage of Gastric Contents Emptied at 1 Hour
Description: Subjects were given a scrambled egg breakfast with toast and a glass of milk. The eggs contained a small amount of a radioactive substance. At the completion of the meal, subjects stood in front of a special camera and pictures were taken at specific intervals. This outcome measure is the proportion of the radiolabeled meal emptied at 1 hour.
Time Frame: Visit 4, approximately 1 hours after radiolabeled meal was ingested
Measure: Median (Inter-Quartile Range); unit: percentage of meal emptied
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
percentage of meal emptied | 12.4 [8 to 18.5] | 38.2 [26.6 to 42.1]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p < .001, ANCOVA

3. Secondary Outcome: Change in Body Weight
Time Frame: baseline, day 30
Measure: Median (Inter-Quartile Range); unit: kg
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
kg | -0.95 [-2.1 to -0.7] | -0.55 [-2.1 to 0.3]
Statistical Analysis 1: Comparison: Exenatide vs Placebo; Test type: Superiority or Other; p = 0.23, ANCOVA

4. Secondary Outcome: Satiation Expressed as Volume to Fullness
Description: In the last 5 days of medication administration, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a visual analog scale (VAS) from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure was the volume consumed when the fullness sensation reached level 3.
Time Frame: Visit 3, approximately 30 minutes after liquid meal
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
mL | 705 [510 to 795] | 675 [413 to 825]

5. Secondary Outcome: Maximum Tolerated Volume
Description: In the last 5 days of medication administration, subjects did a satiation/nutrient drink test. Participants recorded their sensations every 5 minutes using a visual analog scale (VAS) from 0-5, with level 0 being no symptoms, level 3 corresponding to fullness sensation after a typical meal, and level 5 corresponding to the maximal tolerated volume (maximum or unbearable fullness/satiation). This measure was the volume consumed when the fullness sensation reached level 5.
Time Frame: Visit 3, approximately 30 minutes after liquid meal
Measure: Median (Inter-Quartile Range); unit: mL
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
mL | 1244 [918 to 1452] | 1052 [859.1 to 1422]

6. Secondary Outcome: Buffet Meal Intake (kcal)
Description: Five hours after the standard egg meal ingested to measure gastric emptying, subjects were invited to eat, over a 30 minute period, a standard "all you can eat" meal. This meal consisted of either meat or vegetable lasagna, vanilla pudding, and skim milk. Personnel from the study team weighed the food servings post-meal and reported the amount of food left from single portions partially consumed. The total kcal of the food consumed was analyzed by using validated software.
Time Frame: Visit 4, approximately 30 minutes after start of "all you can eat" meal
Measure: Median (Inter-Quartile Range); unit: kcal
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
kcal | 977 [713 to 1336] | 1110 [680.3 to 1658]

7. Secondary Outcome: Aggregate Satiation Symptom Score
Description: Postprandial fullness, nausea, bloating, and pain were measured 30 minutes after the liquid meal using 100 mm horizontal visual analog scales (VAS). The subscale scores could each range from "none"(0) to "worst ever" (100) at the left and right ends of the lines for each symptom. These satiation symptom scores (postprandial fullness, nausea, bloating, and pain) were combined to generate a total scale score with a different total scale range (0 - 400 mm) with 0 mm indicating "none" and 400 indicating "worst ever."
Time Frame: Visit 3, approximately 30 min after ingestion of nutrient drink test
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Exenatide | Placebo
Number analyzed (Participants) | 10 | 10
mm | 145 [133.5 to 204] | 172 [110 to 237]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Exenatide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes